CLINICAL TRIAL: NCT06003283
Title: Tapering of Rituximab Based on Interval Prolongation Compared to Disease Activity-guided Dose Reduction in Patients With Rheumatoid Arthritis: The RITUXERA Trial
Brief Title: Tapering of Rituximab Based on Interval Prolongation Compared to Disease Activity-guided Dose Reduction in Patients With Rheumatoid Arthritis
Acronym: RITUXERA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fonds voor Wetenschappelijk Reumaonderzoek (FWRO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S67309
Record Dates: First submitted 2023-07-19; First posted 2023-08-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Rituximab; Tapering; Disease impact
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Open label multicenter pragmatic randomized controlled superiority trial. Patients will be 1:1 randomized to either the experimental arm or the active comparator arm.
  Study visits are scheduled every 12 weeks (3 months). Recruitment period: 1 year. Trial duration: 2 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tapering of rituximab based on disease activity guided dose reduction (Experimental): Treatment with rituximab every 6 months (24 weeks) with dosing based on disease activity, measured by the DAS28-CRP.
  DAS28-CRP ≤ 3.2: dose reduction according to the following sequence: 1 x 1000 mg IV (maximum), 1 x 500 mg IV, 1 x 200 mg IV (minimum).
  DAS28-CRP > 3.2: administration of previously effective dose.
  Interventions: Drug: Rituximab
- Tapering of rituximab based on interval prolongation (Active Comparator): Treatment with fixed dose of rituximab (1 x 1000 mg IV) if DAS28-CRP ≥ 3.2 AND interval of at least 6 months (24 weeks) since previous administration of rituximab.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — IV rituximab
  Other Names: MabThera; Truxima; Ruxience; Rixathon

SUMMARY:
The goal of this open label multicenter randomized controlled pragmatic superiority trial is to investigate the optimal treatment/tapering strategy with rituximab for patients with rheumatoid arthritis.

The main questions it aims to answer are:

* What is the optimal treatment/tapering strategy for rituximab in patients with rheumatoid arthritis in terms of reducing patient reported disease impact?
* What is the optimal treatment/tapering strategy for rituximab in patients with rheumatoid arthritis in terms of therapeutic efficacy?

Participants will be randomized to one of two study arms:

* Tapering based on disease-activity guided dose reduction (experimental arm)
* Tapering based on interval prolongation (active comparator arm)

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent and participate in the study before any study procedure.
* Age ≥ 18 years.
* Understanding and able to write in Dutch or French.
* Diagnosis of rheumatoid arthritis according to the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Classification Criteria for rheumatoid arthritis.
* Previous response to rituximab, defined as a minimum of one successful rituximab cycle (= a moderate/good EULAR response 16 weeks after the first administration of rituximab).
* Current treatment with rituximab.
* Need for a subsequent rituximab cycle according to the Belgian reimbursement criteria for the use of rituximab in rheumatoid arthritis (DAS28 score ≥3.2).
* Stable dose of methotrexate or other conventional synthetic disease-modifying antirheumatic drugs (DMARDs) 4 weeks prior to baseline.

Exclusion Criteria:

* Current treatment with another biological DMARD than rituximab.
* Current treatment with a targeted synthetic DMARD.
* Pregnancy or pregnancy wish.
* Presence of an absolute contraindication to treatment with rituximab, according to the label of rituximab and according to medical judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of disease impact in both study arms, measured using the Rheumatoid Arthritis Impact of Disease (RAID) questionnaire | Over 2 years (104 weeks)
  RAID questionnaire score range: 0 - 10, with higher scores indicating worse status.

SECONDARY OUTCOMES:
Comparison of disease activity in both study arms, measured using the Disease Activity Score in 28 joints - C-reactive protein (DAS28-CRP) | Over 2 years (104 weeks)
  Main secondary outcome. DAS28-CRP range: 0 - ..., with higher values indicating higher disease activity.
Comparison of disease activity in both study arms, measured using the Simplified Disease Activity Index (SDAI) | Over 2 years (104 weeks)
  SDAI range: 0 - ..., with higher values indicating higher disease activity.
Comparison of cumulative dose of rituximab in both study arms | Over 2 years (104 weeks)
Comparison of cumulative dose of glucocorticoids in both study arms | Over 2 years (104 weeks)
Proportion of patients in both study arms achieving a good or moderate European League Against Rheumatism (EULAR) treatment response after administration of rituximab, over a period of 2 years (104 weeks) | Over 2 years (104 weeks)
  A good EULAR response is defined as a decrease in Disease Activity Score in 28 joints - C-reactive protein (DAS28-CRP) > 1.2 and a present DAS-CRP ≤ 3.2. A moderate EULAR response is defined as a decrease in DAS28-CRP > 0.6 to ≤ 1.2 and a present DAS28-CRP ≤ 5.1, or a decrease in DAS28-CRP > 1.2 and a present DAS28-CRP > 3.2. Treatment responses will be evaluated 12 weeks after every administration of rituximab.
Comparison of loss of disease control in both study arms | Over 2 years (104 weeks)
  Loss of disease control is defined as achieving a Disease Activity Score in 28 joints - C-reactive protein (DAS28-CRP) > 3.2 with previous DAS28-CRP ≤ 3.2.
Comparison of rituximab drug retention rate in both study arms | Over 2 years (104 weeks)
  Defined as the percentage of patients remaining on treatment with rituximab over time.
Proportion of patients tapering rituximab below 1000 mg in the experimental arm | Over 2 years (104 weeks)
Mean/median interval between rituximab administrations in the active comparator group | Over 2 years (104 weeks)
Comparison of serious adverse events/reactions rates in both study arms. | Over 2 years (104 weeks)
  An adverse event or adverse reaction is considered serious if it leads to inpatient hospitalization or prolongation of existing hospitalization, if it results in persistent or significant disability or incapacity, if it results in a life-threatening experience (meaning that the subject was at risk of death), or if it results in death.
Comparison of serious infections rate in both study arms. | Over 2 years (104 weeks)
  An infection is considered serious if it leads to inpatient hospitalization or prolongation of existing hospitalization, if it results in persistent or significant disability or incapacity, if it results in a life-threatening experience (meaning that the subject was at risk of death), or if it results in death.

OTHER OUTCOMES:
Comparison of functional status in both study arms, measured using the Health Assessment Questionnaire - Disability Index (HAQ-DI) | Over 2 years (104 weeks)
  HAQ-DI score range: 0 - 3, with higher scores indicating worse functional status.
Self-efficacy in both study arms, measured using the Arthritis Self-Efficacy Scale (ASES) | Over 2 years (104 weeks)
  ASES score range: 11 - 110, with higher scores indicating higher perceived self-efficacy.
Pain in both study arms, measured using a Visual Analogue Scale (VAS) completed by the patient | Over 2 years (104 weeks)
  VAS pain range: 0 - 100, with higher values indicating higher pain
Fatigue in both study arms, measured using a Visual Analogue Scale (VAS) completed by the patient | Over 2 years (104 weeks)
  VAS fatigue range: 0 - 100, with higher values indicating more fatigue.
Patient global assessment (PGA) of disease in both study arms, measured using a Visual Analogue Scale (VAS) completed by the patient | Over 2 years (104 weeks)
  VAS PGA range: 0 - 100, with higher values indicating worse disease.
Cluster of Differentiation (CD) 19+ and Memory B cell counts in both study arms | Over 2 years (104 weeks)
  Determined at baseline, before administration of rituximab and at year 2 (104 weeks) in both study arms.
Immunoglobulin (Ig) counts (IgG, IgA and IgM) in both study arms | Over 2 years (104 weeks)
  Determined at baseline, before administration of rituximab and at year 2 (104 weeks) in both study arms.
Professional and vocational participation in both study arms, calculated using the Work Productivity and Activity Impairment questionnaire: General Health (WPAI:GH) | Over 2 years (104 weeks)
  The WPAI:GH calculates the percent work time missed due to health (range 0-100, higher numbers indicating more missed work time), the percent impairment while working due to health (range 0-100, higher numbers indicating higher impairment), the percent overall work impairment due to health (range 0-100, higher numbers indicating higher impairment), and the percent activity impairment due to health (range 0-100, higher numbers indicating higher impairment).
Health utility index in both study arms, calculated using the summary index score of the EuroQol - 5 dimensions (EQ-5D) questionnaire | Over 2 years (104 weeks)
  Summary index score range: less than 0 (health state worse than dead, 0 being the value of a health state equivalent to death) to 1 (full health).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Verschueren, MD, PhD, Principal Investigator — University Hospitals Leuven/KU Leuven
Locations (7):
- Belgium (7):
  - ZNA Jan Palfijn, Merksem, Antwerpen
  - Cliniques Universitaires Saint-Luc Bruxelles, Brussels, Brussels Capital
  - Reumacentrum Genk, Genk, Limburg
  - ReumaClinic Genk, Genk, Limburg
  - OLV Aalst, Aalst, Oost-Vlaanderen
  - RZ Heilig Hart, Leuven, Vlaams-Brabant
  - University Hospitals Leuven (UZ Leuven), Leuven, Vlaams-Brabant

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Meyst E, Bertrand D, Joly J, Doumen M, Marchal A, Thelissen M, Neerinckx B, Westhovens R, Verschueren P. Treat-to-target fixed dose rituximab retreatment versus fixed interval retreatment with disease activity-guided rituximab dose optimisation for patients with rheumatoid arthritis: study protocol for a multicentre randomised controlled superiority trial focusing on long-term disease impact (RITUXERA). Trials. 2024 Oct 15;25(1):681. doi: 10.1186/s13063-024-08542-7. PMID 39407334